CLINICAL TRIAL: NCT05693012
Title: Assessment of Early Detection and Prognosis Based on cfDNA Methylation in Myeloma: a Proof of Concept Study
Brief Title: Assessment of Early Detection and Prognosis Based on cfDNA Methylation in Multiple Myeloma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qiu Lugui (Other)
Collaborators: Guangzhou Burning Rock Dx Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Qiu Lugui, Director of lymphoma & myeloma center, Institute of Hematology & Blood Diseases Hospital, China
Organization: Institute of Hematology & Blood Diseases Hospital, China (Other)
Other Study IDs: RSCD2022004
Record Dates: First submitted 2022-12-15; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; early detection; liquid biopsy
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cancer Arm: participants with newly diagnosed multiple myeloma, from whom blood samples will be collected.
  Interventions: Diagnostic Test: cfDNA methylation assessment
- Benign Arm: Participants with newly diagnosed benign hematologic disorders, from whom blood samples will be collected.
  Interventions: Diagnostic Test: cfDNA methylation assessment
- Healthy arm: Participants without known presence of malignancies or certain benign diseases, from whom blood samples will be collected.
  Interventions: Diagnostic Test: cfDNA methylation assessment

INTERVENTIONS:
Diagnostic Test: cfDNA methylation assessment — An exploratory study to establish the early detection and prognosis models of multiple myeloma patients in China based on plasma cf DNA methylation assessment

SUMMARY:
It is an observational, case-control study aimed at early-detection of multiple myeloma and constructing a prognostic model of multiple myeloma. The study will enroll approximately 398 participants including patients with multiple myeloma, patients with benign hematologic disorders and healthy participants.

ELIGIBILITY:
Inclusion Criteria for Cancer Participants:

* Age 40-75 years
* Ability to provide a written informed consent
* Pathologically confirmed diagnosis of multiple myeloma or highly suspicious cases of multiple myeloma
* No prior or ongoing anti-cancer treatment (local or systematic) prior to study blood draw

Inclusion Criteria for Benign Disease Participants:

* Age 40-75 years
* Ability to provide a written informed consent
* Pathologically confirmed diagnosis of benign hematologic disorders or highly suspicious cases with benign hematologic disorders
* No prior or ongoing radical treatment of the benign hematologic disorders prior to study blood draw

Inclusion Criteria for Healthy Participants

* Age 40-75 years
* Ability to provide a written informed consent
* No cancer-related symptoms or other uncomfortable symptoms prior to study blood draw

Exclusion Criteria for All Participants:

* Insufficient qualified blood samples
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant
* Recipient of blood transfusion within 7 days prior to blood draw
* Recipient of anti-tumor drugs to treat non-cancer diseases within 30 days prior to blood draw, such as rheumatic drugs (methotrexate, cyclophosphamide, or azathioprine), or endocrine drugs (tamoxifen)

Additional Exclusion Criteria for Cancer Participants:

• Other current malignant diseases or multiple primary tumors

Additional Exclusion Criteria for Benign Disease Participants:

• Current or history of malignancies

Additional Exclusion Criteria for Healthy Participants:

* Recipient of anti-infectious therapy within 14 days prior to study blood draw
* Prior or ongoing treatment of cancer within 3 years prior to study blood draw
* Current autoimmune disease or clinically significant or uncontrolled comorbidities

Ages: 40 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from the participating medical center and assigned into three arms, including participants with newly diagnosed multiple myeloma, benign hematologic disorders and healthy participants.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of a cfDNA methylation-based early detection modelfor multiple myeloma. | 12 months

SECONDARY OUTCOMES:
The sensitivity and specificity of a cfDNA methylation-based early detection model for multiple myeloma at different clinical stages. | 12 months
The performance of a cfDNA methylation-based prognostic model for multiple myeloma. | 12 months
  Treatment response and survival outcomes, measured by ORR, CR, PFS, and OS, in high-risk group and low-risk group of multiple myeloma.
The specific cfDNA methylation landscape of multiple myeloma in China | 12 months
  The differently methylated regions(DMRs) between multiple myeloma and healthy/benign controls.

CONTACTS AND LOCATIONS:
Overall Officials: Lugui Qiu, MD, Ph.D, Principal Investigator — Chinese Academy of Medical Sciences & Peking Union Medical College
Locations (1):
- National Clinical Research Center for Blood Diseases, Blood Diseases Hospital & Institute of Hematology, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality, China